CLINICAL TRIAL: NCT06818968
Title: A 2-period, Fixed-sequence, Open-label Study to Evaluate the Effect of Multiple Oral Doses of Diltiazem on the Single-dose Pharmacokinetics of MK-6916 in Healthy Participants
Brief Title: A Study of the Effect of Multiple Doses of Diltiazem on the Plasma Levels of MK-6916 in Healthy Participants (MK-6916-005)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 6916-005
Record Dates: First submitted 2025-02-05; First posted 2025-02-11 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Healthy
MeSH Terms: interventions — Diltiazem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MK-6916 + Diltiazem (Experimental): Participants will receive MK-6916 and diltiazem orally.
  Interventions: Drug: MK-6916; Drug: Diltiazem

INTERVENTIONS:
Drug: MK-6916 — Oral administration
Drug: Diltiazem — Oral administration
  Other Names: MK-M793

SUMMARY:
The goal of the study is to learn what happens to levels of MK-6916 in a healthy person's body over time. Researchers will compare what happens to MK-6916 in the body when it is given with or without another medicine called diltiazem.

ELIGIBILITY:
Inclusion Criteria:

The key inclusion criteria include but are not limited to the following:

* Has a body-mass index (BMI) 18 to 32 kg/m^2

Exclusion Criteria:

The key exclusion criteria include but are not limited to the following:

* Has a history of clinically significant endocrine, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or major neurological abnormalities or diseases
* Has a history of cancer (malignancy)
* Has a history of cardiac arrhythmia or recurrent unexplained syncopal events
* Has a first-degree relative with multiple unexplained syncopal events, unexplained cardiac arrest or sudden cardiac death, or has a known family history of an inherited arrhythmia syndrome
* Has positive test(s) for hepatitis B surface antigen, hepatitis C antibodies, or human immunodeficiency virus

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2025-02-27 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-08-08 (Actual)

PRIMARY OUTCOMES:
Area Under the Concentration-Time Curve from Time 0 to Infinity (AUC0-Inf) of MK-6916 | Predose and at designated time points (up to 8 weeks)
  Blood samples will be collected to determine the AUC0-inf of MK-6916.
Area Under the Concentration-Time Curve from Time 0 to 24 hours (AUC0-24hrs) of MK-6916 | Predose and at designated time points (up to 24 hours)
  Blood samples will be collected to determine the AUC0-24 of MK-6916.
Plasma Concentration at 24 Hours (C24) of MK-6916 | Predose and at designated time points (up to 24 hours)
  Blood samples will be collected to determine the C24 of MK-6916.
Plasma Concentration at 12 Hours (C12) of MK-6916 | Predose and at designated time points (up to 12 hours)
  Blood samples will be collected to determine the C12 of MK-6916.
Maximum Plasma Concentration (Cmax) of MK-6916 | Predose and at designated time points (up to 8 weeks)
  Blood samples will be collected to determine the Cmax of MK-6916.
Time to Maximum Plasma Concentration (Tmax) of MK-6916 | Predose and at designated time points (up to 8 weeks)
  Blood samples will be collected to determine the Tmax of MK-6916.
Apparent Clearance (CL/F) of MK-6916 | Predose and at designated time points (up to 8 weeks)
  Blood samples will be collected to determine the CL/F of MK-6916.
Apparent Volume of Distribution (Vz/F) of MK-6916 | Predose and at designated time points (up to 8 weeks)
  Blood samples will be collected to determine the Vz/F of MK-6916.
Apparent Terminal Half-life (t1/2) of MK-6916 | Predose and at designated time points (up to 8 weeks)
  Blood samples will be collected to determine the t1/2 of MK-6916.

SECONDARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 8 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 8 weeks
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The number of participants who discontinue study treatment due to an AE will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (1):
- Fortrea CRU, Madison ( Site 0001), Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com